CLINICAL TRIAL: NCT00265837
Title: Phase III Trial of T Lymphocyte Depletion by Elutriation and CD34 Add-Back for Allogeneic Bone Marrow Transplantation
Brief Title: Laboratory-Treated Donor Bone Marrow in Treating Patients Who Are Undergoing a Donor Bone Marrow Transplant for Hematologic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: J0165 CDR0000454926; P01CA015396 (NIH); P30CA006973 (NIH); JHOC-J0165; JHOC-WIRB-1908; JHOC-WIRB-20020342
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: graft versus host disease; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; childhood acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; chronic myelomonocytic leukemia; juvenile myelomonocytic leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; Philadelphia chromosome negative chronic myelogenous leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult immunoblastic large cell lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Hodgkin Disease; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Therapeutics

INTERVENTIONS:
Biological: graft versus host disease prophylaxis/therapy
Procedure: allogeneic bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor bone marrow transplant or peripheral blood stem cell transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When certain stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Removing the T cells from the donor cells before transplant may stop this from happening.

PURPOSE: This randomized phase III trial is studying donor bone marrow that is treated in the laboratory using two different devices to compare how well they work in treating patients who are undergoing a donor bone marrow transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness, in terms of incidence of graft failure and incidence of greater than grade 1 acute graft-vs-host disease, of ex vivo manipulation of bone marrow cells comprising counterflow centrifugal elutriation for T-lymphocyte depletion followed by CD34-positive stem cell selection using CliniMACS vs Isolex 300i in patients with a hematologic malignancy undergoing allogeneic bone marrow transplantation from an HLA-identical sibling donor.

OUTLINE: This is a randomized study. Patients are stratified by age (< 40 vs 40-65) and disease status (low-risk [i.e., chronic phase chronic myelogenous leukemia, acute myeloid leukemia in first complete remission (CR), acute lymphocytic leukemia in first CR, Hodgkin's or non-Hodgkin's lymphoma in sensitive relapse, or multiple myeloma in CR or partial remission) vs high-risk [i.e., all others]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Allogeneic bone marrow cells are subjected to counterflow centrifugal elutriation (CCE) for T-lymphocyte depletion. The elutriation fractions are then processed over 2-2.5 hours using CliniMACS to select for CD34-positive stem cells.
* Arm II: Allogeneic bone marrow cells are subjected to CCE for T-lymphocyte depletion. The elutriation fractions are then processed over 4-4.5 hours using Isolex 300i to select for CD34-positive stem cells.

Patients in both arms then undergo ex vivo manipulated, T-lymphocyte-depleted, CD34-positive stem cell-selected, allogeneic bone marrow transplantation on day 0.

After the transplantation, patients are followed periodically for 1 year.

PROJECTED ACCRUAL: A total of 206 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies or genetic disorders:

  * Acute myeloid leukemia (AML), meeting 1 of the following criteria

    * Primary resistant disease
    * Disease in complete remission (CR)
    * Disease in first early relapse
    * Secondary AML arising out of myelodysplastic syndrome
  * Acute lymphocytic leukemia (ALL), meeting 1 of the following criteria:

    * Primary resistant disease
    * Disease in CR
    * Disease in first early relapse
  * Chronic myelogenous leukemia
  * Myelodysplastic syndrome (MDS)
  * Chronic myelomonocytic leukemia
  * Philadelphia chromosome-negative myeloproliferative disorder
  * Multiple myeloma
  * Hodgkin's lymphoma
  * Non-Hodgkin's lymphoma
  * Genetic disorders or inborn errors of metabolism
* Planning allogeneic bone marrow transplantation at the Sidney Kimmel Comprehensive Cancer Center at the Johns Hopkins Medical Center

  * Must have an HLA-identical sibling donor by serologic or molecular typing of HLA class I antigens and molecular typing of HLA class II antigens

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior red blood cell or platelet transfusion from the same donor

Other

* Concurrent participation in another clinical trial allowed

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2002-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Incidence of graft-vs-host disease or graft failure

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Jones, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States